CLINICAL TRIAL: NCT07179458
Title: Word Retrieval in Aphasia
Brief Title: Criterion-learning Naming Treatment For Addressing Comprehension Deficits in Aphasia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Thomas Jefferson University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Erica Middleton, Institute Scientist, Jefferson Moss Rehabilitation Research Institute, Albert Einstein Healthcare Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4526.4; R01DC015516 (NIH)
Record Dates: First submitted 2025-08-25; First posted 2025-09-17 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Aphasia
Keywords: anomia; retrieval practice; word-finding problem; communication disorder; naming impairment; word comprehension impairment
MeSH Terms: conditions — Aphasia; Anomia; Communication Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Criterion-learning practice (Experimental): This is a single-arm study
  Interventions: Behavioral: Criterion-learning practice

INTERVENTIONS:
Behavioral: Criterion-learning practice — The experiments will be presented on a computer. On each criterion-learning trial, a picture is presented and the participant is asked to try to produce the name for the object with or without a cue. Correct-answer feedback is provided. Criterion learning involves presenting a block of items in fixed order, and on each trial, the experimenter or a voice-recognition component will code the response during the trial as correct/incorrect. When the item reaches its assigned criterion level, it is dropped from further training in a session.

SUMMARY:
Aphasia is a disorder of spoken and written language, most commonly following a stroke. It is estimated that between 2.5 and 4 million Americans are living with aphasia today. A common problem in aphasia involves difficulty retrieving known words in the course of language production and comprehension. The overarching goal of this project is to develop and test early efficacy, efficiency, and the tolerability of a lexical treatment for aphasia in multiple-session regimens that are comprised of retrieval practice, distributed practice, and training dedicated to the elicitation of correct retrievals. The aim of this work is to add to and refine the evidence base for the implementation and optimization of these elements in the treatment of production and comprehension deficits in aphasia, and make important steps towards an ultimate goal of self-administered lexical treatment grounded in retrieval practice principles (RPP) to supplement traditional speech-language therapy that is appropriate for People with Aphasia (PWA) from a broad level of severity of lexical processing deficit in naming and/or comprehension. This project cumulatively builds on prior work to develop a theory of learning for lexical processing impairment in aphasia that aims to ultimately explain why and for whom familiar lexical treatments work, and how to maximize the benefits they confer.

DETAILED DESCRIPTION:
This study examines a retrieval practice-based naming treatment termed criterion learning. In criterion learning, each item's assigned criterion level dictates the number of times that item is correctly retrieved before it is dropped from further training within a session. Criterion learning optimally incorporates potent learning experiences, including spaced retrieval practice with emphasis on correct retrievals during training. The present study will provide critical observations for optimizing criterion learning for treating word processing deficits in people with aphasia. This study will recruit 20 community-dwelling individuals with aphasia, who will undergo comprehensive neuropsychological characterization. Subsequently, participants will engage in an experimental treatment designed to promote improvements in word processing deficits.

This study will examine transfer from two types of naming treatment to word comprehension performance. Each PWA will perform naming treatment in one session at different dosages with a test of comprehension performance administered approximately one week and one month following treatment. Main outcomes of interest will be degree of transfer of each type of naming treatment to comprehension performance.

ELIGIBILITY:
Inclusion Criteria:

* English as a native or primary language
* Adults with stroke who are at least 6 months post-onset
* Exhibit semantic comprehension deficit, defined as a minimum of 80 errors on word-picture verification pre-test

Exclusion Criteria:

* History of comorbid neurological diagnoses, such as Multiple Sclerosis or Parkinson's Disease
* History of a learning disability that significantly impacted language development, such as developmental language disorder
* Insufficient stamina to participate in the protocol

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Trained comprehension items | approximately one-week and one-month following treatment
  Word-picture verification task

SECONDARY OUTCOMES:
Trained naming items | a single session held during a single day, scheduled at the participant's convenience but typically held within two weeks following pre-treatment assessment
  Confrontation naming task that involves trained items
Trained comprehension items | pre-treatment
  Word-picture verification task
Untrained comprehension items | pre-treatment, approximately one-week and one-month post-treatment
  Word-picture verification task

CONTACTS AND LOCATIONS:
Overall Officials: Erica L Middleton, PhD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Jefferson Moss Rehabilitation Research Institute, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data and analysis code will be accessible on the Open Science Framework (OSF).
Supporting Information: Analytic Code
Time Frame: 6 months following publication
Access Criteria: Anonymized data and analysis code will be accessible on the Open Science Framework (OSF).

DOCUMENTS (1):
  • Informed Consent Form (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT07179458/ICF_001.pdf